CLINICAL TRIAL: NCT02503475
Title: Stanford Center for Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Redlich Professor Departments of Anesthesiology, Perioperative and Pain Medicine | Neurosciences | Neurology (by courtesy), Chief, Division of Pain Medicine, Director, Stanford Systems Neuroscience and Pain Lab (SNAPL), Stanford University, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22436
Record Dates: First submitted 2015-07-15; First posted 2015-07-21 (Estimated); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Project 1- Real-Time fMRI (Other): This arm investigates Real-Time fMRI within 4 groups:
  Attention Regulation (AR) Group- Experimental Cognitive Regulation (CR) Group- Experimental Sham Group- Sham Comparator Free Strategy Group- Active Comparator
  Interventions: Other: Real-Time fMRI
- Project 2 - CBT/MBSR (Experimental): This arm investigates 2 experimental groups:
  Cognitive Behavioral Therapy (CBT) Mindfulness Based Stress Reduction (MBSR)
  Interventions: Behavioral: CBT or MBSR
- Project 3- Acupuncture (Other): This arm investigates Acupuncture within 2 groups:
  Verum- Experimental Sham- Sham comparator
  Interventions: Device: Acupuncture

INTERVENTIONS:
Other: Real-Time fMRI — Real-Time fMRI: AR, CR, Sham, and Free Strategy groups will be compared to determine the following:
  (1) whether a cognitive strategy improves rtfMRI neurofeedback to modulate brain activity and pain; (2) which strategy is most effective at individual and group levels at modulating brain activity and pain; and (3) whether the investigators can predict individual ability to modulate brain activity or pain using a particular strategy and applying mixed effects modeling of treatment efficacy using baseline measurements.
  Arms: Project 1- Real-Time fMRI
Behavioral: CBT or MBSR — CBT/MBSR: The study will investigate whether CBT versus MBSR differentially enhance behavioral and neural indices of the ability to implement cognitive regulation (CR) and attention regulation (AR) during evoked pain in the lower back in participants with chronic low back pain. An additional wait list control (WL) group will be used to determine the effects of time on pain symptom severity and well-being.
  Arms: Project 2 - CBT/MBSR
Device: Acupuncture — Acupuncture: The investigators will compare the efficacy and mechanisms of verum and sham electroacupuncture.
  Arms: Project 3- Acupuncture

SUMMARY:
The purpose of the Stanford Center for Back Pain is to investigate and characterize the mechanisms of four treatments for chronic low back pain. These interventions (research treatment) include real-time fMRI neurofeedback, mindfulness based stress reduction, cognitive behavioral therapy, and acupuncture treatment. The investigators plan to characterize both mechanisms of treatment effects and efficacy.

DETAILED DESCRIPTION:
The Stanford Center for Back Pain establishes a collaborative, multidisciplinary research program to investigate CAM interventions for the treatment of chronic low back pain (CLBP). The investigators' overall goal is to characterize the shared and distinct mechanisms of four CAM interventions and translate the investigators' findings to tailored and effective treatments for CLBP. CLBP is a highly prevalent and difficult-to-treat condition for which many patients seek CAM therapies. Basic science has revealed that abnormalities in central pain modulatory and emotion regulatory systems play a crucial role in CLBP. What is not clear is how CAM therapies alter the functioning of the brain systems involved in chronic pain. The Stanford Center for Back Pain aims to fill this gap by conducting 3 projects, each aiming at elucidating mechanisms underlying different CAM therapies for CLBP.

Project 1 will focus on a promising novel alternative therapy for CLBP real-time fMRI neurofeedback which trains patients to control specific neural processes that lead to improvements in pain. Project 2 will characterize the pain modulatory and emotion regulatory effects of mindfulness based stress reduction and cognitive behavioral therapy for CLBP. Project 3 will characterize psychophysical and neuroimaging based neural mechanisms underlying verum and placebo acupuncture.

The Stanford Center for Back Pain will provide optimal collaboration and synergy within a multidisciplinary framework to identify mechanisms of CAM therapies for CLBP so that they can eventually translate them into enhance clinical care of CLBP.

ELIGIBILITY:
Inclusion Criteria:

* English Fluency
* Chronic Low Back Pain as defined by NIH task-force or Healthy Controls

Exclusion Criteria:

* MRI contraindications
* Pregnant or planning to become pregnant
* Medical conditions that would interfere with study procedures, at the discretion of the study team
* Neurologic disorder, history of seizures, stroke, or brain abnormalities, which would interfere with brain integrity, at the discretion of the study team.
* Mental health conditions or treatment for mental health problems that would interfere with study procedures, at the discretion of the study team.
* Other project specific criteria may apply.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in pain severity | Up to 12 months post-treatment
  Visual Analogue Scale from 0 to 100, where 0=no pain and 100=worst pain imaginable

SECONDARY OUTCOMES:
Changes in pain symptom severity and well being | Up to 12 months post-treatment
  Responses to NIH PROMIS measures such as Pain Interference, Pain Behavior, Physical Function, Fatigue, Sleep Disturbance

CONTACTS AND LOCATIONS:
Overall Officials: Sean Mackey, MD, PhD, Principal Investigator — Stanford University; James Gross, PhD, Principal Investigator — Stanford University; Rachel Manber, PhD, Principal Investigator — Stanford University; Sean Mackey, MD, PhD, Study Director — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Derived] Karayannis NV, Smuck M, Law C, Mackey SC, Gross JJ, Darnall BD, Hush J. Self-reported physical function is strongly related to pain behavior and pain interference and weakly related to physical capacity in people with chronic low back pain. Musculoskelet Sci Pract. 2023 Feb;63:102721. doi: 10.1016/j.msksp.2023.102721. Epub 2023 Jan 23. PMID 36759316
- [Derived] Mackey S, Gilam G, Darnall B, Goldin P, Kong JT, Law C, Heirich M, Karayannis N, Kao MC, Tian L, Manber R, Gross J. Mindfulness-Based Stress Reduction, Cognitive Behavioral Therapy, and Acupuncture in Chronic Low Back Pain: Protocol for Two Linked Randomized Controlled Trials. JMIR Res Protoc. 2022 Sep 27;11(9):e37823. doi: 10.2196/37823. PMID 36166279
- [Derived] Kong JT, MacIsaac B, Cogan R, Ng A, Law CSW, Helms J, Schnyer R, Karayannis NV, Kao MC, Tian L, Darnall BD, Gross JJ, Mackey S, Manber R. Central mechanisms of real and sham electroacupuncture in the treatment of chronic low back pain: study protocol for a randomized, placebo-controlled clinical trial. Trials. 2018 Dec 13;19(1):685. doi: 10.1186/s13063-018-3044-2. PMID 30541586